CLINICAL TRIAL: NCT03172637
Title: Female Sexual Dysfunctions in Patients With Chronic Renal Failure
Brief Title: Female Sexual Dysfunction in Renal Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Esraa Ahmed Mohamed (Other)
Responsible Party: Sponsor-Investigator, Esraa Ahmed Mohamed, GP, Assiut University
Organization: Assiut University (Other)
Other Study IDs: FSDRF
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Evaluations of Sexual Dysfunction of Female in Chronic Renal Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: 50 female end stage renal disease patients
- Group B: 50 normal female patients

SUMMARY:
A myriad of sexual problems affect men and women with chronic kidney disease (CKD), including decreased libido, erectile dysfunction, dysmenorrhea, and infertility. Menstrual abnormalities are common in CKD and many women are an-ovulatory .

Causes of sexual dysfunction in CKD include hormonal alterations along with vascular, neurologic, psychogenic, and other factors, such as medications, contribute to the development of sexual dysfunction . Sexual dysfunction in females is mainly due to hormonal factors and manifests mainly as menstrual irregularities, amenorrhea, lack of vaginal lubrication, and failure to conceive.

DETAILED DESCRIPTION:
Hormonal changes in chronic kidney disease are seen in prolactine, gonadotropins, and gonadal hormones. In women with CKD, elevated levels of follicle-stimulating hormone (FSH) and luteinizing hormone (LH) are common. These hormonal changes are detected in the early stages of kidney disease and progressively worsen as kidney disease progresse .

. Women with chronic renal failure commonly have elevated circulating prolactin levels. As in men with chronic renal failure, the hypersecretion of prolactin in this setting appears to be autonomous, as it is resistant to maneuvers designed to stimulate or inhibit its release.

It has been suggested that the elevated prolactin levels may impair hypothalamic-pituitary function and contribute to sexual dysfunction and galactorrhea in these patients. However, uremic women treated with bromocryptine rarely resume normal menses and continue to complain of galactorrhea (if present), despite normalization of the plasma prolactin concentration. Thus, factors other than hyperprolactinemia must be important in this setting .

ELIGIBILITY:
Inclusion Criteria:

* -Female patients with chronic renal failure (eGFR <15 ml/min/1.7m2 ) on dialysis or not.
* Age from 18 to 45 years old.
* Married.
* Sexually active during the last 6 monthes.

Exclusion Criteria:

* Pregnant women.
* Other medical diseases ( diabetes mellitus ,cardiac disorders ,neurological disorders and other systematic diseases).
* Taking medications affect sexuality function e.g. antidepressant drugs.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: The Female Sexual Function Index (FSFI) will be used to assess sexual function .This index includes 19 questions related to 6 parameters: sexual desire, sexual arousal, lubrication, orgasm, sexual satisfaction and dyspareunia. A face-to-face inter-view with each participant in which the FSFI questions will be verbally asked and answered and compare between them in effect of renal failure on sexuality.
  Duration of chronic renal failure duration of dialysis ,number of sessions of dialysis per week,medical treatment, haemoglobin and creatinine level will be fullfilled.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
effect of chronic renal failure in females on their sexuality function | two years
  compare sexuality function between female with chronic renal failure and normal female and observe difference between two groups